CLINICAL TRIAL: NCT04822025
Title: A Phase II, Prospective, Randomized, Double-Blind, Dose-Comparison, Multi-Center Study to Evaluate the Safety, Tolerability, and Immunogenicity of the SARS-CoV-2 Vaccine Candidate MVC-COV1901 in Elderly Adults
Brief Title: A Study to Evaluate MVC-COV1901 Vaccine Against COVID-19 in Elderly Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medigen Vaccine Biologics Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CT-COV-23
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2021-06

CONDITIONS: Covid19 Vaccine
Keywords: Covid19 vaccine
MeSH Terms: interventions — MVC-COV1901 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Dose (Experimental): High-Dose S-2P protein with CpG and Aluminum Hydroxide/0.5mL
  Interventions: Biological: MVC-COV1901 (High-Dose)
- Mid Dose (Experimental): Mid-Dose S-2P protein with CpG and Aluminum Hydroxide/0.5mL
  Interventions: Biological: MVC-COV1901(Mid-Dose)

INTERVENTIONS:
Biological: MVC-COV1901 (High-Dose) — Approximately 300 participants will receive 2 doses of MVC-COV1901(S-2P protein with adjuvant) at Visit 2 (Day 1) and Visit 4 (Day 29) via intramuscular (IM) injection in the deltoid region
  Arms: High Dose
Biological: MVC-COV1901(Mid-Dose) — Approximately 100 participants will receive 2 doses of MVC-COV1901(S-2P protein with adjuvant) at Visit 2 (Day 1) and Visit 4 (Day 29) via intramuscular (IM) injection in the deltoid region
  Arms: Mid Dose

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of MVC-COV1901 vaccine in two different dose forms in participants who are generally healthy or with stable pre-existing health conditions.

DETAILED DESCRIPTION:
This is a Phase II, prospective, randomized, double-blinded (investigator/site staff and participants; Sponsor open), dose-comparison, multi-center study. Participants who are generally healthy or with stable pre-existing health conditions will be randomized, stratified by comorbidity. All eligible participants will be randomized to receive 2 doses of either High-dose or Mid-dose of MVC-COV190 in a predefined ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant ≥ 65 years of age at randomization.
2. Healthy adults or adults with pre-existing medical conditions who are in stable condition. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease 3 months before enrollment and expected to remain stable for the duration of the study.
3. Participant is willing and able to comply with all required study visits and follow-up required by this protocol.
4. Participant has not travelled overseas within 14 days of screening and will not have any oversea traveling throughout the study period.
5. Participant is able to understand and comply with study requirements/procedures (if applicable, with assistance by caregiver, surrogate, or legally authorized representative) based on the assessment of the investigator and must provide written informed consent.

Exclusion Criteria:

1. Employees at the investigator's site, of the Sponsor or the contract research organization (CRO) who are directly involved in the conduct of the study.
2. Currently receiving or received any investigational intervention within 30 days prior to the first dose of study intervention.
3. Administered any licensed live-attenuated vaccines within 28 days or other licensed non-live-attenuated vaccines within 7 days prior to the first dose of study intervention.
4. Administered any blood product or intravenous (IV) immunoglobulin administration within 12 weeks prior to the first dose of study intervention.
5. Participant previously received any coronavirus vaccine.
6. Currently receiving or anticipate to receive concomitant immunosuppressive or immune-modifying therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or < 2 weeks of daily receipt of prednisone less than 20 mg or equivalent) within 12 weeks prior to the first dose of study intervention.
7. Currently receiving or anticipate to receive treatment with tumor necrosis factor (TNF)-α inhibitors, e.g. infliximab, adalimumab, etanercept within 12 weeks prior to the first dose of study intervention.
8. Major surgery or any radiation therapy within 12 weeks prior to the first dose of study intervention.
9. Immunosuppressive illness or immunodeficient state, including hematologic malignancy, history of solid organ, bone marrow transplantation, or asplenia.
10. A history of malignancy with potential risk for recurrence after curative treatment, or current diagnosis of or treatment for cancer (exceptions are squamous and basal cell carcinomas of the skin and treated uterine cervical carcinoma in situ, at the discretion of the investigator).
11. Bleeding disorder considered a contraindication to intramuscular injection or phlebotomy.
12. Participant with known human immunodeficiency virus (HIV) infection or who is HIV antibody positive, with CD4 count < 350 cells/mm3 or a detectable HIV viral load within the past year (low level variations from 50-500 viral copies/mL or equivalent which do not lead to changes in antiretroviral therapy [ART] are permitted).
13. Participant who, in the investigator's judgement, is not in stable condition and by participating in the study could adversely affect the safety of the participant, interfere with adherence to study requirements or evaluation of any study endpoint. This may include aparticipant with ongoing acute diseases, severe infections, autoimmune disease, laboratory abnormality or serious medical conditions in the following systems: cardiovascular, pulmonary, hepatic, neurologic, metabolic, renal, or psychiatric.
14. Participant with previous known SARS-CoV-1 or 2 infection or potential exposure to SARS-CoV-1 or 2 viruses (EXCEPT for those who have been tested negative or completed the self-managements/ home quarantines/ home isolations)
15. Participant with a history of hypersensitivity to any vaccine or a history of allergic disease or reactions likely to be exacerbated by any component of the MVC-COV1901.
16. Body (oral, rectal, or ear) temperature ≥ 38.0°C or acute illness (not including minor illnesses such as diarrhea or mild upper respiratory tract infection at the discretion of the investigator) within 2 days before the first dose of study intervention.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 420 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events(AEs) [Safety and Tolerability] | Day 1 to 28 days after the second vaccination
  To evaluate the incidence of Adverse Events(AEs) of MVC-COV1901 from Visit 2 (Day 1) to Visit 6 (28 days after the second dose of study intervention) in terms of the number and percentage of participants with the occurrence of:
  Solicited local AEs (up to 7 days after each dose of study intervention) Solicited systemic AEs (up to 7 days after each dose of study intervention) Unsolicited AEs (up to 28 days after each dose of study intervention) AE of Special Interest (AESI) Vaccine-Associated Enhanced Disease(VAED) Serious adverse events (SAEs)
Immunogenicity of MVC-COV1901 | Day 1 to 28 days after the second vaccination
  To evaluate the immunogenicity of High-dose MVC-COV1901, as compared to Mid-dose MVC-COV1901, in terms of neutralizing antibody titers.

SECONDARY OUTCOMES:
Incidence of Adverse Events(AEs) [Safety and Tolerability] | Day 1 to 180 days after the second vaccination
  To evaluate the Incidence of Adverse Events(AEs) of MVC-COV1901 over the study period in terms of the number and percentage of participants with the occurrence of:
  >= Grade 3 AE AE of Special Interest (AESI) Vaccine-Associated Enhanced Disease(VAED) Serious adverse events (SAEs)
Immunogenicity of MVC-COV1901 | Day 1 to 180 days after the second vaccination
  The antigen-specific immunoglobulin titers and neutralizing antibody titers at Visit 4 (28 days after the first dose of study intervention), Visit 6 (28 days after the second dose of study intervention), Visit 7 (90 days after the second dose of study intervention) and Visit 8 (180 days after the second dose of study intervention) in terms of antigen-specific immunoglobulin titers and neutralizing antibody titers

CONTACTS AND LOCATIONS:
Overall Officials: Szu-Min Hsieh, MD, Principal Investigator — National Taiwan University Hospital; Tzou-Yien Lin, MD, Principal Investigator — Chang Gang Memorial Hospital, LinKou
Locations (4):
- Taiwan (4):
  - Hualien Tzu Chi Hospital, Hualien City
  - Shuang H Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Hospital Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Waits A, Chen JY, Cheng WH, Yeh JI, Hsieh SM, Chen C, Janssen R, Lien CE, Lin TY. Safety and immunogenicity of MVC-COV1901 vaccine in older adults: Phase 2 randomized dose-comparison trial. Int J Infect Dis. 2022 Nov;124:21-26. doi: 10.1016/j.ijid.2022.08.021. Epub 2022 Aug 29. PMID 36049700